CLINICAL TRIAL: NCT05553834
Title: A Phase II Study of PCSK9 Inhibitor Alirocumab and PD-1 Inhibitor Cemiplimab in Patients With Metastatic, Refractory To Prior Anti PD-1 Non-small Cell Lung Cancer: TOP2201
Brief Title: PCSK9 Inhibitor and PD-1 Inhibitor in Patients With Metastatic, Refractory To Prior Anti PD-1 Non-small Cell Lung
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00111111
Record Dates: First submitted 2022-09-02; First posted 2022-09-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-08

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — alirocumab; cemiplimab

STUDY DESIGN:
Intervention Model Description: Combination therapy involving anti-PCSK9 antibody alirocumab with the anti-PD-1 antibody cemiplimab.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Alirocumab and Cemiplimab (Experimental): Combination of anti-PCSK9 antibody alirocumab with the anti-PD-1 antibody cemiplimab
  Interventions: Combination Product: Alirocumab and Cemiplimab

INTERVENTIONS:
Combination Product: Alirocumab and Cemiplimab — Combination of PCSK9 inhibitor Alirocumab 150mg SC q2weeks and PD-I inhibitor Cemiplimab 350mg IV q3 weeks

SUMMARY:
PCSK9 mediates immune checkpoint blockade resistance by downregulating tumor cell surface MHC class 1 molecules. This study will evaluate if combining the anti-PCSK9 antibody alirocumab with the anti-PD-1 antibody cemiplimab can generate anti-tumor activity and clinical responses in patients with metastatic lung cancer who have progressed on first line immune checkpoint blockade therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented recurrent and/or metastatic non-small cell lung cancer
* Progression after prior PD-1 directed therapy (as monotherapy or in combination with chemotherapy and/or anti-CTLA4, or anti-VEGF agents) - defined as investigator assessed progression from prior treatment
* If molecularly altered NSCLC including EGFR, ALK, ROS1, MET exon 14, RET, BRAF, NTRK, progression on prior targeted therapy is required
* Measurable disease by RECIST 1.1
* ECOG Performance Status 0 or 1
* Signed written informed consent
* Minimum of 4 weeks from any other experimental anti-cancer therapies or prior PD-1 treatment
* Meet all the laboratory criteria per protocol

Exclusion Criteria:

* Prior treatment with PCSK9 inhibitors
* Cardiac issues including MI, uncontrolled arrhythmia, symptomatic angina pectoris, active ischemia, or cardiac failure not controlled by medications.
* Uncontrolled diabetes mellitus, defined as HbA1c > 10
* Major surgery less than 4 weeks prior to study enrollment
* Another malignant condition diagnosed within 3 years of study enrollment
* Intolerance to prior PD-1/L1 treatment including discontinuation for severe or recurrent severe toxicity (including myocarditis or other myocardiotoxity, encephalitis, colitis, diarrhea, pancreatitis, hypo/hyperthyroidism, hypopituitarism, adrenal insufficiency, rash, autonomic neuropathy, myasthenia gravis, Guillain-Barre, myositis/polymyositis, hepatitis, Type 1 Diabetes, thrombocytopenia) or developed an immune checkpoint blockade related immune adverse event that was refractory to steroids and required additional systemic immunosuppressive medication.
* Known history of HIV seropositivity or known acquired immunodeficiency syndrome (AIDS)
* Additional exclusion criterion as per listed in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-16 (Actual); Primary Completion 2025-09-16 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Response rate associated with combination of alirocumab and cemiplimab | Day 1 of treatment until the date of first documented progression or date of death, whichever comes first, assessed up to 110 weeks per RECIST 1.1
  Ascertain the response rate associated with alirocumab and cemiplimab, with 95% confidence intervals. Response rate is defined as the proportion of treated subjects with a complete or partial response per RECIST 1.1 criteria. All patients who receive at least one dose of alirocumab and cemiplimab will be considered for the primary outcome analysis

SECONDARY OUTCOMES:
Safety and tolerability of the combination regimen | Day 1 of treatment until 30 days post last dose
  Toxicity analysis will be performed on a continual basis following CTC V 5.0 criteria
Progression Free Survival | Day 1 of treatment until the date of first documented progression or date of death, whichever comes first, assessed up to 110 weeks
  Progression Free Survival will be assessed utilizing RECIST 1.1 criteria
Overall survival | Day 1 of treatment until death or off study due to any other reason whichever comes first, assessed up to 110 weeks
  Patients will be followed till death or off study due to any other reason

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Moffitt Cancer Center, Tampa, Florida
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No